CLINICAL TRIAL: NCT04381923
Title: High Flow Nasal Oxygen Versus Continuous Positive Airway Pressure Helmet Evaluation: A Randomized Crossover Trial in COVID-19 Pneumonia
Brief Title: COVIDNOCHE Trial (HFNO Versus CPAP Helmet) in COVID-19 Pneumonia
Acronym: COVIDNOCHE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain IRB approval
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Timothy Gaulton, M.D., Assistant Professor of Anesthesiology and Critical Care, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 843124
Record Dates: First submitted 2020-05-07; First posted 2020-05-11 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2; Hypoxemic Respiratory Failure; Pneumonia, Viral; COVID
MeSH Terms: conditions — Respiratory Insufficiency; Pneumonia, Viral

STUDY DESIGN:
Intervention Model Description: This will be a randomized study with alternating treatment assignment in which all advanced respiratory units will be assigned to use one of two default interventions (helmet CPAP vs HFNO) as the first-line treatment for refractory hypoxemia (defined as an oxygen saturation (Sp02) of 92% or less on on ≥ 6 LPM (liters per minute) nasal cannula (NC) oxygen). The first-line treatment will be alternated in each unit at 14-day intervals. The initial assignment will be determined by a computer randomization scheme. Patients who are still on their assigned intervention during crossover will remain on that assigned intervention. A design with numerous short periods and frequent crossovers was selected to minimize the risk of changes over time in the patient population and usual care confounding trial results. A 14-day period is also felt to be the minimal time needed to ensure device availability and adherence.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Helmet Continuous Positive Airway Pressure (CPAP) (Active Comparator): When a patient has an Sp02 < 92% on ≥ 6 LPM NC, helmet CPAP will be applied unless a specific contraindication is present.
  Interventions: Device: Helmet Continuous Positive Airway Pressure (CPAP)
- High Flow Nasal Oxygen (HFNO) (Active Comparator): When a patient has an Sp02 < 92% on ≥ 6 LPM NC , HFNO (≥ 40 LPM) will be applied unless a specific contraindication is present
  Interventions: Device: High Flow Nasal Oxygen (HFNO)

INTERVENTIONS:
Device: Helmet Continuous Positive Airway Pressure (CPAP) — Helmet CPAP will be initiated at a pressure of 5 cmH20 and fraction of inspired oxygen (Fi02) of < 60%. If oxygen saturation (Sp02) remains < 92%, pressure will be increased to 10 cmH20. FiO2 will then be tapered to target a SpO2 ≥ 92%. Breaks with intervening HFNO use will be provided as needed for meals and during hours of sleep.
  Arms: Helmet Continuous Positive Airway Pressure (CPAP)
Device: High Flow Nasal Oxygen (HFNO) — HFNO will be initiated at a flow rate of 40 LPM and a fraction of inspired oxygen (Fi02) of < 60%. If oxygen saturation (SpO2) remains < 92%, the flow rate will be increased to 60 LPM. FiO2 will then be adjusted to target a SpO2 ≥ 92%. Patients with discomfort due to HFNO may have their flow rate decreased until the discomfort resolves.
  Other Names: High Flow Nasal Cannula (HFNC)
  Arms: High Flow Nasal Oxygen (HFNO)

SUMMARY:
The purpose of the COVIDNOCHE trial (HFNO versus CPAP Helmet Evaluation in COVID-19 Pneumonia) is to evaluate the comparative effectiveness of standard care non-invasive respiratory support (helmet CPAP versus HFNO) for acute hypoxemic respiratory failure from COVID-19 pneumonia on ventilator-free days (primary outcome) and other clinical outcomes measured up to 90 days.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is a respiratory illness that can cause acute arterial hypoxemia. Treatment with invasive ventilation improves oxygenation yet results in death in over 50% of cases. The high incidence of disease has also reduced resources needed to safely deliver invasive ventilation including mechanical ventilators and intravenous sedation. Non-invasive respiratory support has been shown to be efficacious in acute hypoxemic respiratory failure from other etiologies and has the potential to reduce rates of intubation and the time spent on mechanical ventilation in COVID-19. However, it is unknown which type of support is the most effective, limiting the ability to improve clinical outcomes and appropriately allocate resources. To help guide clinical practice and policy, it is critical to understand the comparative effectiveness of two forms of non-invasive respiratory support used worldwide, continuous positive airway pressure (CPAP) delivered via a helmet interface and high flow nasal oxygen (HFNO).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with confirmed COVID-19 with an Sp02 < 92% on ≥ 6 liters NC admitted to a Penn Medicine advanced respiratory unit. An advanced respiratory unit is a unit capable of non-invasive respiratory support such as an ICU or intermediate care unit.

Exclusion Criteria:

Patients will be excluded if they meet ≥ 1 of the following criteria based on current Penn Medicine respiratory guidelines and prior trials of non-invasive respiratory support:

* Respiratory failure related to other etiology (e.g. exacerbation of chronic obstructive pulmonary disease, acute pulmonary edema)
* Baseline oxygen requirement
* Diagnosis of acute or chronic hypoventilation
* Tracheostomy
* Claustrophobia
* Prior intubation during hospitalization
* Urgent need for endotracheal intubation
* Other contraindications to non-invasive respiratory support (glasgow coma scale lower than 8, absence of airway protective gag reflex, elevated intracranial pressure, upper airway obstruction)
* Patient dose not wave to receive the assigned intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Ventilator-Free Days (VFD) | 28 days
  VFD is the number of days alive and free of mechanical ventilation in the first 28 days after study enrollment. Death before 28 days will be assigned a VFD equal to 0 to penalize non-survival. In cases of repeated intubation and extubation, periods free from invasive ventilation and lasting at least 24 consecutive hours will be calculated and summed. Timing of intubation and extubation will be captured in hours, and the number of hours a patient received invasive ventilation will be used to calculate duration of ventilation.

SECONDARY OUTCOMES:
ICU and Hospital Length of Stay | 28 days
  Days spent in the ICU and hospital after time of enrollment
Intubation | 28 days
  Incidence and time to intubation in days after the time of enrollment
Renal Replacement Therapy (RRT) | 28 days
  Incidence of RRT after the time of enrollment
Mortality | 28 days, 90 days
  Death from any cause during after the time of enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States